CLINICAL TRIAL: NCT05128201
Title: Consolidative Radiotherapy Combined With Camrelizumab and Chemotherapy for Oligometastatic Nasopharyngeal Carcinoma: A Multicenter, Open-Label, Phase II Trial (NPC-CR01)
Brief Title: Consolidative Radiotherapy Combined With Camrelizumab and Chemotherapy for Oligometastatic Nasopharyngeal Carcinoma
Acronym: NPC-CR01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-CR01; 2020-PT320-004 (Other Grant/Funding Number: NHC Key Laboratory of NPC)
Record Dates: First submitted 2021-11-06; First posted 2021-11-19 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Oligometastatic Disease
Keywords: local consolidative radiotherapy; oligometastatic nasopharyngeal carcinoma; Progression-free survival; immune checkpoint inhibitor

STUDY DESIGN:
Intervention Model Description: System chemotherapy (Camrelizumab , Gemcitabine and cisplatin or nedaplatin) And local consolidative radiotherapy for all metastatic lesion, and Maintenance of Camrelizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- System treatment plus consolidative radiotherapy and Maintenance treatment (Experimental): 4-6 Cycles System chemotherapy (Camrelizumab , Gemcitabine and cisplatin or nedaplatin) ; And local consolidative radiotherapy for all metastatic lesion (30-45Gy/3-8F) and Maintenance of Camrelizumab (total 2 years; from first cycles of System chemotherapy to last cycles of miantenance of camrelizumab)
  Interventions: Radiation: consolidative radiotherapy

INTERVENTIONS:
Radiation: consolidative radiotherapy — local consolidative radiotherapy for all metastatic lesion (30-45Gy/3-8F)
  Other Names: local consolidative radiotherapy

SUMMARY:
The purpose of this study is to explore the efficacy and tolerance of local consolidative radiotherapy combined with Camrelizumab and chemotherapy in patients with oligometastatic nasopharyngeal carcinoma

DETAILED DESCRIPTION:
This trial was a single-arm, multicenter phase Ⅱ clinical study. Eligible oligometastatic NPC patients were scheduled to evaluate the efficacy and tolerance of local consolidative radiotherapy combined with camrelizumab and chemotherapy in patients with oligometastatic NPC. Progression-free survival (PFS) determined will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-70 years old, no gender limit;
* 2. Oligo metastasis is defined as less than or equal to 5 metastatic lesions and less than or equal to 2 metastatic organs
* 3. Patients with an ECOG score of 0 or 1, and an expected survival period of ≥6 months;
* 4. Has good organ function:

  1. Hematology: WBC>3.0×109/L; ANC>1.5×109/L; Hb>90g/L; PLT>100×109/L; Albumin ≥3g/dL;
  2. Liver function: bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with known Gilbert disease and serum bilirubin level ≤ 3 times ULN can be included), AST and ALT ≤ 3 times ULN (if liver metastases occur , Then AST/ALT≤5 times ULN), and alkaline phosphatase≤3 times ULN (if liver or bone metastasis occurs, ALP≤5 times ULN); （3） Coagulation function: International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; （4）Renal function: According to the Cockcroft-Gault formula (Appendix 8), serum creatinine ≤1.5 times ULN or creatinine clearance ≥60mL/min.
* 5. Female subjects have a negative pregnancy test (for female patients with fertility); female patients without fertility;
* 6. Male patients with fertility and female patients with fertility and risk of pregnancy must agree to take adequate contraceptive measures throughout the study period, and contraception lasts for 12 months after receiving this program.
* 7. Patients who are willing and able to comply with visit arrangements, treatment plans, laboratory tests and other research procedures;
* 8. During the research period, they are willing to comply with the arrangement and cannot participate in any other clinical research on drugs and medical devices;
* 9. For patients who have previously received neoadjuvant chemotherapy, adjuvant chemotherapy, radiotherapy or radiotherapy for non-metastatic diseases, the time from the last chemotherapy and/or radiotherapy to randomization must reach a non-treatment interval of ≥ 6 months . Oral S1 and capecitabine have no requirement for treatment interval for those who are progressing during chemotherapy.
* 10. The patients sign a formal informed consent form to show that they understand that this study complies with the hospital's policies

Exclusion Criteria:

* 1. Those who have a history of severe immediate hypersensitivity to any of the drugs used in this study;
* 2. Suffered from other malignant tumors other than nasopharyngeal carcinoma within 5 years (except for tumors with an expected 5-year OS>90%, such as non-melanoma skin cancer or pre-invasive cervical cancer);
* 3. Any of the following conditions in the 6 months before screening: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient cerebral ischemia Onset or symptomatic pulmonary embolism. Patients with known coronary artery disease, congestive heart failure that does not meet the above criteria, or left ventricular ejection fraction <50% must adopt an optimized and stable medical plan determined by the treating doctor. If appropriate, you can consult a cardiologist;
* 4. Have received any of the following treatments:

  1. Have received anti-PD-1 or anti-PD-L1 antibody therapy in the past;
  2. Have received any investigational drug within 4 weeks before using the investigational drug for the first time;
  3. A large number of glucocorticoids or other immunosuppressants (including but not limited to prednisone, dexamethasone, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor) have been used in the 4 weeks before treatment Subjects with anti-TNF drugs, or subjects in need of hormone therapy during clinical trials. Other special circumstances require communication with the sponsor. In the absence of active autoimmune diseases, inhaled or topical steroids and adrenal cortex hormones with a dose> 10 mg/day of prednisone are allowed to be substituted;
  4. Those who have been vaccinated with anti-tumor vaccines or the study drug has been vaccinated with live vaccines within 4 weeks before the first administration;
  5. Have undergone major surgery or severe trauma within 4 weeks before using the study drug for the first time;
  6. Enroll in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up;
* 5. Patients with active autoimmune disease or a history of autoimmune disease but may relapse. Remarks: Patients with the following diseases are not excluded and can enter further screening:

  1. Controlled type 1 diabetes
  2. Hypothyroidism (if only hormone replacement therapy can be used to control)
  3. Skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, hair loss)
  4. Any other diseases that are not expected to recur without external triggers
* 6. Active infections, including tuberculosis, hepatitis B, hepatitis C and human immunodeficiency virus. Patients with positive HBV surface antigen (HBsAg) but HBV DNA <1000 copies/mL are eligible to participate in this study; patients with positive HCV antibody test results are only allowed if the HCV RNA polymerase chain reaction test results are negative. Be selected for this study;
* 7. Idiopathic pulmonary fibrosis, drug-induced pneumonia, organizing pneumonia (bronchiolitis obliterans), idiopathic pneumonia, or chest CT scan at the time of screening shows evidence of active pneumonia;
* 8. Drug abuse or alcohol addiction;
* 9. No capacity for civil conduct or limited capacity for civil conduct;
* 10. The patient has a physical or mental illness, and the researcher believes that the patient cannot fully or fully understand the possible complications of this study;
* 11. Other serious acute or chronic medical conditions (including immune colitis, inflammatory diseases, Enteropathy, non-infectious pneumonia, pulmonary fibrosis) or mental illness (including dementia and epilepsy, recent, past year or active suicidal ideation or behavior) or abnormal laboratory tests;
* 12. Patients whose expected survival time is less than 6 months;
* 13. Patients with significantly reduced heart, liver, lung, kidney and bone marrow functions
* 14. Previously diagnosed as immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related diseases;
* 15. Female patients during pregnancy or lactation, male or female patients who are fertile but are unwilling or unable to use contraception during the entire study period and at least one year after the end of the treatment plan;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The time from the start of treatment to the first observation of disease progression or death from any cause (whichever occurs first)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  the proportion of patients achieving the optimal overall remission (complete or partial remission)
Disease control rate (DCR) | 2 years
  the proportion of patients with the best efficacy (CR or PR or SD)
Overall survival (OS) | 3 years
  the time from the start of treatment to death from any cause
Duration of Overall Response (DOR) | 2 years
  the time the patient first reaches complete or partial remission to disease progression

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No
After completing the treatment plan, we will report our research plan and research results.